CLINICAL TRIAL: NCT00200213
Title: The Effect of Portion Size and Quantity of Food Provided on Intake
Brief Title: Liking of Snack Foods - Sub-Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2107-02
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Eating Behavior; Obesity; Satiation
MeSH Terms: conditions — Feeding Behavior; Obesity

INTERVENTIONS:
Behavioral: portion or unportioned food

SUMMARY:
Specific Aims: Environmental factors contributing to overconsumption, such as larger food portion sizes, may be contributing to the obesity epidemic. The objective of the proposed study is to examine the independent and combined effects of portion size and quantity of food on intake in normal weight males and females. Participants will be randomly assigned to one of four conditions varying in the portion size and quantity of junk food provided: small quantity of food packaged in small portions (SSP), small quantity of food packaged in large portions (SLP), large quantity of food packaged in small portions (LSP), and large quantity of food packaged in large portions (LLP). A box containing four different junk foods, packaged according to one of the four conditions, will be given to participants to take home for three days. The total amount of food consumed from the box over the three days will be measured. It is anticipated that portion size and quantity of food, both independently and combined, will influence intake, such that larger portion sizes and quantity of food provided to participants will produce greater intake.Subject Population: We propose to recruit 60 healthy men and women, aged 18-50 years, with a body mass index (BMI) of less than or equal to 28. Participants will be non-smokers, unrestrained eaters, and have no known food allergies to the foods used in the investigation.Methods/Design: Participants will be randomly assigned to one of four conditions, varying in portion size (small versus large) and quantity of food provided (small versus large). A box containing four junk foods, packaged according to one of the conditions, will be provided to participants. They will be encouraged to eat as much or as little of the food as they want, but to at least taste each of the four foods over the three-day period. During this time, they will be instructed to not eat any other junk foods. At the end of the three-day period, participants will return the box with any remaining uneaten junk food.Data Analyses: The dependent variables, the amount of grams and kcals consumed from the provided junk foods, will be examined between the four different conditions.Significance: If portion size and quantity are related to intake, subsequent studies will develop clinical interventions related to reducing portion size and/or quantity of food available in the household.

ELIGIBILITY:
Inclusion Criteria:

Healthy, non-smoking, normal- and over-weight (body mass index [BMI] < 30) unrestrained, males and females, who regularly eat junk foods (consume junk foods > 3 times per week).

Exclusion Criteria:

Participants will be excluded if they are not between the ages of 18 and 50, smoke, following a weight loss diet, an athlete in training, pregnant or breastfeeding, or have a health condition or use medication that affects eating or requires specialized diet therapy (e.g., diabetes). Additionally, if participants rarely consume junk foods (< 2 times per week) or have allergies or unfavorable preferences towards foods used in the investigation they will be excluded from the study. Participants will also be excluded if they are a restrained eater (scoring > 12 on the Three Factor Eating Questionnaire [TFEQ] [Stunkard & Messick, 1985]) or report being a binge eater.-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32
Dates: Start 2004-02; Study Completion 2005-03

PRIMARY OUTCOMES:
Amount of food eaten

SECONDARY OUTCOMES:
Liking of foods in study

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Weight Control and Diabetes Research Center, Providence, Rhode Island, United States